CLINICAL TRIAL: NCT02857127
Title: Promoting Physical Activity for Vulnerable Adults and Elderly People: Evaluation of a Walking Program in Primary Care Settings
Brief Title: Physical Activity Promotion in Primary Health Care Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Grace Angélica de Oliveira Gomes, Doctor, Universidade Federal de Sao Carlos
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FAPESP14/03909-2
Record Dates: First submitted 2016-07-30; First posted 2016-08-05 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Motor Activity
Keywords: Low income population; Motor Activity; Primary Health Care
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Group (Experimental): A group of people who participated in the walking program during a six month period. This group also received an educational material and attended meetings for behavioral change strategies.
  Interventions: Behavioral: Walking program
- Control Group (No Intervention): A group of people who did not receive the educational material and did not participated in any of the activities offered by the research team, such as walking classes and meetings for behavioral change.

INTERVENTIONS:
Behavioral: Walking program — To encourage people to exercise more through a behavioural and educational intervention during six months and other six months of follow up.
  Arms: Intervention Group

SUMMARY:
A quasi experimental study evaluating the effectiveness of a walking program at primary health care settings in a low-income area

DETAILED DESCRIPTION:
There is a high prevalence of physical inactivity (AF) in the world and in Brazil. Offering programs of physical activity becomes a convenient option to increase the physical activity level of the population and promote aging process more active and healthy over the life. There is need for greater depth in relation to the operation of programs to promote physical activity and the effects of these programs on different biopsychosocial aspects, especially those offered in primary care settings. This research aims to evaluate a walking program geared to adults and seniors on the following aspects:

1. Characteristics and operation of the intervention,
2. effects of behavior change to physical activity, and
3. biopsychosocial effects of physical activity.

It is a quasi experimental and controlled study, with: 1) intervention group (n = 71), 2) and control group (n = 71). The intervention will last for six months, with a subsequent follow-up period of six months after the intervention. The program will offer supervised exercise twice a week, lasting an hour. The classes will consist of recreational activities, walking and educational strategies of behavior change for physical activity. Variables will be evaluated for attendance, barriers to physical activity, waiver reasons, physical activity level, sociodemographic, socioeconomic and biopsychosocial aspects. Most females, aged over 40 years, low levels of education, income and varied biopsychosocial characteristics are expected. After the intervention, it is expected that the program present characteristics of low adhesion and retention, especially because of the barrier "lack of time". Still, the promotion of supervised walking increase levels of physical activity beyond the time provided by the program and it will improve the biopsychosocial conditions of the participants.

ELIGIBILITY:
Inclusion Criteria:

* To be insufficiently active
* To accept the intervention invitation
* Living around the selected primary health care
* To sign the Term os Consent
* To have 18 years or more

Exclusion Criteria:

* To participate only in one day of intervention
* To have less than 75% of presence in the intervention
* To give up of the intervention

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Subjective evaluation of physical activity level evaluated through the International Physical Activity Questionnaire | six months
  Physical activity level evaluated through the International Physical Activity Questionnaire
Objective evaluation of physical activity level evaluated through accelerometer device | six months
  Physical activity level evaluated through accelerometer device

CONTACTS AND LOCATIONS:
Overall Officials: Grace AO Gomes, Doctor, Principal Investigator — Universidade Federal de Sao Carlos
Locations (1):
- Secretaria Municipal de Saúde, São Carlos, São Paulo, Brazil

REFERENCES:
- [Derived] Baba CT, Oliveira IM, Silva AEF, Vieira LM, Cerri NC, Florindo AA, de Oliveira Gomes GA. Evaluating the impact of a walking program in a disadvantaged area: using the RE-AIM framework by mixed methods. BMC Public Health. 2017 Sep 15;17(1):709. doi: 10.1186/s12889-017-4698-5. PMID 28915827